CLINICAL TRIAL: NCT07134712
Title: Safety and Efficacy Study of Intravenous Administration of MiSaver (Umbilical Cord Blood Derived Nucleated Cells) After Acute Myocardial Infarction
Brief Title: Safety and Efficacy of MiSaver (CB Cells) for Acute Myocardial Infarction, Phase II
Acronym: SEMIAMI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HONYA Medical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CshKmuhHcmmh2024; CS1-24127 (Other: The Institutional Review Board Chung Shan Medical University Hospital); 24CT053Ae (Other: MacKay Memorial Hospital Institutional Review Board Approval of Clinical Trial); KMUHIRB-F(I)-20250025 (Other: Kaohsiung Medical University Chung-Ho Memorial Hospital Institutional Review Board)
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: heart attack; stem cell; Cardiovascular diseases
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LDRSB (Experimental): One-time infusion 0.5 x10^7 TNCs/kg
  Interventions: Biological: Cord Blood Nucleated cells
- MDRSB (Experimental): One-time infusion 1.6 x10^7 TNCs/kg
  Interventions: Biological: Cord Blood Nucleated cells
- PCRSB (Placebo Comparator): One-time infusion saline 30ml
  Interventions: Biological: Cord Blood Nucleated cells

INTERVENTIONS:
Biological: Cord Blood Nucleated cells — MiSaver will be administered via peripheral intravenous injection. Based on dosage, the experimental group will be divided into two subgroups: 0.5 × 10⁷ or 1.6 × 10⁷ nucleated cells per kilogram of patient body weight.

SUMMARY:
This trial is a Phase II, multicenter clinical study. The purpose of this trial is to evaluate the safety and efficacy of MiSaver, a cellular therapy product, in patients who have experienced an acute myocardial infarction (AMI). Specifically, the study aims to assess the improvement in left ventricular function of the heart following the administration of MiSaver, as well as to determine the safety of using stem cell therapy in these patients.

This trial will employ a single-blind design (subject-blinded), meaning that the participants will not be aware of whether they are receiving MiSaver or standard treatment, while the researchers will have this information. This design helps ensure transparency and adherence to ethical standards while also providing valuable clinical insights.

By utilizing randomization, we can enhance the reliability and comparability of the study results. A portion of the participants will receive MiSaver, while the others will undergo standard treatment. This allows for a direct comparison of the two therapeutic approaches to determine their respective efficacy.

The primary objective of this trial is to evaluate the safety and efficacy of MiSaver, in the treatment of patients with acute myocardial infarction (AMI). To achieve this, we will collect comprehensive participant data, including assessments of cardiac function, records of cardiac events, and quality-of-life surveys. By analyzing these data, we aim to gain a deeper understanding of the benefits and limitations of this treatment approach.

DETAILED DESCRIPTION:
We will enroll patients who have been diagnosed with acute myocardial infarction (AMI) within a timeframe of 36 hours to 7 days after the initial diagnosis. Eligible participants must be hemodynamically stable at the time of enrollment. Hemodynamic stability is defined as not requiring vasopressor support within the past 24 hours, having a systolic blood pressure (SBP) of less than 80 mmHg for no more than one hour, and not experiencing a resting heart rate of over 100 beats per minute for more than one hour.

Additionally, eligible patients must have undergone successful reperfusion therapy or coronary angiography confirming the absence of infarction at the time of screening. Only patients who are willing to receive MiSaver cellular therapy will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years, BMI ≤ 32
2. Patients diagnosed with acute myocardial infarction by a cardiologist, within 36 hours to 7 days post-diagnosis, and able to complete cell infusion within this period.
3. Left ventricular ejection fraction (LVEF) ≤ 45%, hemodynamically stable patients who do not require vasopressor support within 24 hours.
4. Patients with a history of coronary artery disease, who have previously undergone percutaneous coronary intervention or coronary artery bypass graft surgery, may also be included upon evaluation by a cardiologist.
5. Patients deemed unsuitable for percutaneous coronary intervention or coronary artery bypass graft surgery by a cardiologist.
6. Must agree to sign the informed consent form.
7. Subjects must use effective contraception during the study observation period and for 6 months after its conclusion to ensure no pregnancy occurs during the study. (Primarily for women of childbearing potential).
8. Agree to and comply with the required outpatient visits and examinations during the study observation period.

Exclusion Criteria:

1. Age < 45 years, BMI > 32.
2. Women who are planning to become pregnant, are pregnant, or are breastfeeding
3. Immunodeficiency diseases caused by infection , such as Human Immunodeficiency Virus (HIV).
4. Patients diagnosed as needing coronary artery bypass surgery or potentially requiring coronary revascularization surgery within the next 6 months.
5. Severe aortic or mitral valve stenosis.
6. Life-threatening arrhythmias.
7. Malignant tumors, including all categories and cancer conditions.
8. Hematologic disorders or other severe organ diseases with an expected survival of less than one year.
9. Chronic kidney disease (eGFR < 30 mL/min/1.73m²) or patients undergoing dialysis.
10. Patients with autoimmune diseases or those who have already received immunotherapy.
11. Patients who have undergone tumor treatment or require immunosuppressive therapy within the last three years.
12. History of transfusion reactions.
13. Recipients of bone marrow or organ transplants.
14. Liver dysfunction (bilirubin > 2.5 mg/dL or transaminases > 5x the upper limit of normal).
15. Patients who have previously received growth factors, cytokines, gene therapy, or stem cell therapy.
16. Subjects participating in more than one clinical trial.
17. Inability to sign the consent form or comply with outpatient follow-up after infusion therapy.
18. Patients with a known allergy to this product or its excipients (e.g., dimethyl sulfoxide, cell preservation solution).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AE | From enrollment to the end of treatment at 12 months
  Collection and assessment of all adverse events within 12 months after treatment, including type, incidence, and severity.
GVHD | at the 3rd month after infusion.
  Proportion of patients developing Graft Versus Host Disease (GVHD) at the 3rd month after infusion.
cardiovascular composite events | From enrollment to the end of treatment at 12 months.
  Number and frequency of cardiovascular composite events, including myocardial infarction and stroke.

SECONDARY OUTCOMES:
LVEF | Cardiac function was evaluated with 2D Doppler echo before treatement and at the third, sixth, ninth and 12th month.
  Evaluation of treatment efficacy through 2D echocardiography to assess left ventricular volume and ejection fraction.
Cardiovascular-related mortality | 12 months after treatment
  Cardiovascular-related mortality record within 12 months after treatment
Incidence of new myocardial infarction (NMI) | 12 months after treatment
  Incidence of new myocardial infarction (NMI), with a clear definition provided, such as symptoms, elevated cardiac enzymes, and ECG changes.
  d. Non-fatal stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Kwo-Chang Ueng, PhD, Study Director — Chung Shan Medical University
Locations (3):
- Taiwan (3):
  - Mackay Memorial Hospital Hsinchu Branch, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital Daqing Branch, Taichung

IPD SHARING:
Plan to Share IPD: Undecided